CLINICAL TRIAL: NCT06013722
Title: Strategy for Unstable Coronary Plaque in Patients Presenting to the Emergency Department for Chest Pain Suspected of Coronary Artery Disease. A Trial in Primary Prevention and Cardiovascular Risks Evaluation
Brief Title: Strategy for Unstable Coronary Plaque in Patients Presenting to Emergency Department for Chest Pain Suspected of Coronary Artery Disease
Acronym: SPECTRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Monaco Scientific center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-CHITS-007
Record Dates: First submitted 2023-07-29; First posted 2023-08-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerosis
Keywords: Atherosclerotic plaques; Acute coronary syndrome; 18F-Na PET; Coronary Artery Calcification Score
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients of groups III and IV (Experimental): Patients who are categorized after calcium score determination as presenting an intermediate risk to produce atheromatous plaques (group III : between the 40th percentile and the 65th percentile) or presenting a high risk to produce such plaques (group IV: >65th percentile).
  Interventions: Diagnostic Test: 18F-Na PET Scan

INTERVENTIONS:
Diagnostic Test: 18F-Na PET Scan — For the intermediate risk population who would demonstrate within 6 to 18 months after first calcium score either an increase of percentile of more than 20% or an increase above 20 points of the calcium score and for high risk population, 18F-Na PET scan will be recommended and repeated 6 months later. Secondary prevention treatment will then be administered in the event of an abnormal examination.

SUMMARY:
Primary prevention of coronary disease and especially its major complication, inaugural myocardial infarction, is based on any prodromal symptoms identification and on risk profile establishment. About 50% of myocardial infarctions are caused by an unstable non-stenosing plaque, asymptomatic before the event since without significant reduction in coronary flow, particularly during a stress test or during stress imaging.

Study purpose is to set up, in medical emergency department, check-up unit and cardiology department, a primary prevention strategy articulated around a routine examination: calcium scoring. The latter makes it possible to categorize patients according to their risk of generating atheromatous plaques and to classify them into several risk levels (groups) according to their score: low (<40th percentile), intermediate (between the 40th percentile and the 65th percentile: group III) or high risk (>65th percentile, group IV). 18F-Na PET scan can mark unstable coronary plaques. For the intermediate risk population who would demonstrate within 6 to 18 months after first calcium score either an increase of percentile of more than 20% or an increase above 20 points of the calcium score and for high risk population, 18F-Na PET scan will be recommended and repeated 6 months later. Secondary prevention treatment will then be administered in the event of an abnormal examination.

DETAILED DESCRIPTION:
The purpose of this protocol is to determine the frequency and the mapping of unstable coronary plaques highlighted by 18F-Na PET in patients at intermediate and high risk, as well as their evolution under treatment.

Aside from traditional risk factors collection and related biological assessments, risk establishment is based on calcium score, a simple non-injected and very little irradiating scanner which measures coronary calcifications, stigmata of healed atheroma plaques and, as a rule, non-evolving. Calcium score, which is interpreted according to age, sex and ethnicity, therefore makes it possible to assign a percentile within the distribution of all the patients and to classify patients in:

* Group I: "absence of atheromatous plaques": Score 0
* Group II: patients generating few plaques (low risk): calcium score above zero and classifying the patient below the 40th percentile of a similar population;
* Group III: patients generating moderate plaques (intermediate risk) with a calcium score classifying the patient equal or above the 40th percentile and less than the 65th percentile;
* Group IV: patients generating a lot of plaques (high risk): calcium score classifying the patient equal or above the 65th percentile. These are more likely to be patients who will come from the cardiology / check-up sector because of a higher probability of symptoms or of already being treated for primary prevention.

Study assumptions are:

* apart from any hemodynamically significant coronary stenosis, the instability of a plaque can lead to symptomatic but transient micro-thrombotic phenomena which are spontaneously (or under the effect of an anti-aggregation/anticoagulation) resorbable. Regardless of this plaque fate (most frequently scarring, with calcifications, or much more rarely inaugural acute coronary syndrome and therefore infarction), it is a major coronary event which must switch the patient from primary prevention to secondary prevention;
* on painful thoracic syndromes that are sufficiently suggestive to require immediately to rule out an acute coronary syndrome or secondarily myocardial ischemia (angina), identifying a rapid progression of the coronary involvement (on the basis of calcium score) or the direct demonstration of plaque instability (by 18F-Na coupled with a CT scan) is a major cardiovascular prevention endpoint;
* in patients consulting for this clinical presentation, determining the frequency of those with rapid coronary evolution and/or instability of coronary plaque(s) represents a fundamental preliminary epidemiological study to modify prevention approach of primary coronary artery disease;
* the evaluation by non-invasive coronary imaging of secondary prevention treatment impact on these same patients initially diagnosed as "rapidly progressive" and/or unstable would make it possible to consolidate this strategy if it proves to be effective on the basis of plaque images and clinical follow-up (in terms of events).

ELIGIBILITY:
Inclusion Criteria:

* Patient with no coronary history presenting to the emergency room, to the assessment unit or having consulted in the cardiology department for suspicious chest pain that does not allow an acute coronary syndrome or angina to be excluded and:

  * in whom the diagnosis of acute coronary syndrome has been ruled out on the basis of clinical, electrocardiographic, biological monitoring, or even by imaging (including coronary angiography), in accordance with recommendations and good practices
  * in whom effort myocardial ischemia is rendered unlikely on the basis of a clinical and paraclinical evaluation (either ergometric or by functional imaging: scintigraphy, echography or stress MRI)
  * wishing diagnostic care and primary prevention of coronary disease.
* Age above or equal to 18 and strictly below 80 years old
* Having given informed consent

Exclusion Criteria:

* Pregnant woman
* Patient with cognitive disorders
* Claustrophobic patient, or refusing radiological examinations
* Patient refusing cardiological follow-up and/or treatment of his risk factors or refusing to participate in the study
* Patient with contraindications or intolerances to HMG-CoA reductase inhibitors (statins) and/or Ezetimibe
* Patient with liver failure
* Patient with myopathy or with a history of (rhabdo)myolysis
* Marked arrhythmia and in particular supraventricular or ventricular hyperexcitability, or chronic or paroxysmal atrial fibrillation not controlled by antiarrhythmic treatment
* Patients with a history of sternotomy or valve replacement or metallic intracardiac probes, generators of scanner artefacts
* Calcium score corresponding to the percentiles of groups I and II
* For patients in groups III and IV:

  * renal insufficiency with glomerular filtration rate estimated by the MDRD and/or CKD-EPI formula less than or equal to 55 ml/min/1.73 m2,
  * known intolerance to radiological contrast products, or in whom an injected CT scan has already been performed in the 6 months preceding inclusion
* Person participating in another biomedical research
* Person under judicial protection (guardianship, curatorship...)
* Person deprived of liberty by a judicial or administrative decision.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Unstable coronary plaque evolution description through calcium score variation | 8 months
  Unstable coronary plaque evolution will be described through calcium score variation calculation.
Unstable coronary plaque evolution description through coro-scanner plaque size variations | 8 months
  Unstable coronary plaque evolution will be described through coro-scanner plaque size variations measurement
Unstable coronary plaque evolution description through coro-scanner plaque density variations | 8 months
  Unstable coronary plaque evolution will be described through coro-scanner plaque density variations measurement
Unstable coronary plaque evolution description through coro-scanner morphological aspect variations | 8 months
  Unstable coronary plaque evolution will be described through coro-scanner morphological aspect variations
Unstable coronary plaque evolution description through coro-scanner variations in terms of stenosis diameter | 8 months
  Unstable coronary plaque evolution will be described through coro-scanner variations in terms of stenosis diameter
Unstable coronary plaque evolution description through 18F-Na PET scan target binding variations | 8 months
  Unstable coronary plaque evolution will be described through 18F-Na PET scan binding variations (number of targets).
Unstable coronary plaque evolution description through 18F-Na PET scan binding intensity variations | 8 months
  Unstable coronary plaque evolution will be described through 18F-Na PET scan binding variations (SUVmax for each target).

SECONDARY OUTCOMES:
Effectiveness of primary cardiovascular prevention strategy initiation by the care team | 24 months
  Evaluation at study end of the number of patients having entered the monitoring system, the number of patients with signs of coronary involvement and percentage of patients with coronary progression criteria.
Comparison of study cohort symptoms evolution to the symptoms evolution of an historical local cohort with comparable symptomatology which motivated the implementation of a "secondary prevention type" treatment | 24 months
  The number of persistent symptoms increasing and leading to the prescription of new tests (based on clinical management and good practices) and the number of symptoms having completely disappeared will be compared between the study cohort and the local historical one.
Compare, between study cohort and historical cohort, the rate of occurrence of cardiovascular events of interest | 24 months
  Number of following cardiovascular events will be presented:
  * angina proved by biology, ECG and functional and/or anatomical imaging,
  * coronary revascularization in the territory of the unstable plaque if it is individualized or any revascularization (angioplasty or bypass),
  * myocardial infarction,
  * occurrence of a ventricular arrhythmia,
  * cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick CLAESSENS, MD-PhD, Study Director — Centre Hospitalier Princesse Grace
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No